CLINICAL TRIAL: NCT00382096
Title: A Randomized, Double-blind, Active-controlled, Multicenter Study to Compare the Effect of 24 Weeks Treatment With a Fixed Combination Therapy of Vildagliptin and Metformin to the Individual Monotherapy Components in Drug Naive Patients With Type 2 Diabetes
Brief Title: Efficacy of Fixed Combination Therapy of Vildagliptin and Metformin Compared to the Individual Monotherapy Components in Drug Naive Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLMF237A2302
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; metformin; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Vildagliptin + Metformin Dose 1 (Experimental)
  Interventions: Drug: Vildagliptin + Metformin
- Vildagliptin + Metformin Dose 2 (Experimental)
  Interventions: Drug: Vildagliptin + Metformin
- Vildagliptin (Active Comparator)
  Interventions: Drug: Vildagliptin
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin
Drug: Metformin
  Arms: Metformin
Drug: Vildagliptin + Metformin
  Arms: Vildagliptin + Metformin Dose 1; Vildagliptin + Metformin Dose 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a fixed combination of vildagliptin and metformin in lowering blood glucose in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female (non-fertile or of childbearing potential using a medically approved birth control method) patients with type 2 diabetes
* Diagnosis of T2DM for at least 4 weeks prior to study entry
* Age 18 - 78 years inclusive
* Body mass index (BMI) of 22 - 40 kg/m2
* HbA1c: 7.5 - 11% inclusive
* FPG <270 mg/dL (15 mmol/L)

Exclusion Criteria

* Pregnant or lactating female
* A history of type 1 diabetes
* Evidence of significant diabetic complications
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06-03 (Actual); Study Completion 2008-06-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | At week 24

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | At week 24
Percent of patients with endpoint HbA1c <7% | At week 24
Percent of patients with reduction in HbA1c >/=0.7% | At week 24
Adverse event profile after treatment | At week 24
Change from baseline in body weight | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Multiple Locations, Germany

REFERENCES:
- See also: Clinical Trial Results for CLMF237A2302 at Novartis Clinical Trials.com — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2650